CLINICAL TRIAL: NCT01332331
Title: A Randomized, Open Label Study Comparing Safety and Efficacy Parameters for a High and a Low Dose of Ambrisentan (Adjusted for Body Weight) for the Treatment of Pulmonary Arterial Hypertension in Paediatric Patients Aged 8 Years up to 18 Years
Brief Title: Efficacy and Safety of Ambrisentan in Children 8-18yrs
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ongoing juvenile rat toxicology studies.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112529; 2010-019547-19 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-04-11 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary arterial hypertension; pediatric
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose Ambrisentan (Experimental): body weight 20 to 35 kg - 2.5 mg; body weight 35 kg and over - 5.0 mg
  Interventions: Drug: Ambrisentan - low dose
- High Dose Ambrisentan (Experimental): body weight 20 to 35 kg - 5.0 mg; body weight 35 to 50 kg - 7.5 mg; body weight 50 kg and over - 10.0 mg
  Interventions: Drug: Ambrisentan - high dose

INTERVENTIONS:
Drug: Ambrisentan - low dose — body weight 20 to 35 kg - 2.5 mg; body weight 35 kg and over - 5.0 mg
  Arms: Low Dose Ambrisentan
Drug: Ambrisentan - high dose — body weight 20 to 35 kg - 5.0 mg; body weight 35 to 50 kg - 7.5 mg; body weight 50 kg and over - 10.0 mg
  Arms: High Dose Ambrisentan

SUMMARY:
A 6-month (24-week), randomized, open label evaluation of the safety, tolerability, and efficacy of a high and low dose ambrisentan (adjusted for body weight) treatment group in subjects aged 8 years up to 18 years with pulmonary arterial hypertension (PAH). An additional objective is to determine the ambrisentan population pharmacokinetics in the paediatric population. The study will include a screening/baseline period and a treatment period. The treatment period will be 24 weeks or until the subject's clinical condition deteriorates to the point that alternative/additional treatment is necessary. Patients who participate in the study and in whom continued treatment with ambrisentan is desired will be eligible to enrol into a long term follow-up study. The primary comparison will be the safety and tolerability of the two ambrisentan dose groups (Low vs. High) in the paediatric PAH population The secondary comparison will be the change from baseline for the efficacy parameters between the two treatment groups.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare, progressive, highly debilitating disease characterized by vascular obstruction and the variable presence of vasoconstriction, leading to increased pulmonary vascular resistance and right-sided heart failure. If left untreated, PAH ultimately leads to right ventricular failure and death; adult subjects have a median survival of 2.8 years without treatment. Epidemiological estimates vary but prevalence in Europe is thought to be of the order of 15 cases per million. Large scale epidemiology studies of PAH in children have not been conducted and there is no or limited outcome data in pediatric PAH patients. A register in France (1995-1996) estimates the prevalence in children is as low as 3.7 cases per million. In a national, comprehensive country wide survey of the epidemiology of idiopathic PAH (IPAH) management and survival in the United Kingdom (UK) the incidence was 0.48 cases per million children per year and the prevalence was 2.1 cases per million children.

Ambrisentan (VOLIBRIS™ tablets) is an endothelin receptor antagonist (ERA) marketed in the European Union (EU) and some other countries by GlaxoSmithKline (GSK) and in the United States as LETAIRIS® by Gilead Sciences Inc. Ambrisentan is indicated for the treatment of adult patients with PAH to improve exercise capacity, decrease the symptoms of PAH, and delay clinical worsening.

The primary purpose of this paediatric study is to provide clinically relevant information on the safety and pharmacokinetic profile of ambrisentan in children with the most common causes of PAH in this age group. The design of the study is also intended to provide information to guide dose selection and supportive efficacy data in this age group. Despite the fact that none of the currently available adult treatments are licensed for use in children <12 yrs, (with the exception of bosentan which was recently approved for use in paediatric population from 2 years of age) they are widely used off label. This study will provide useful prescribing information to the medical community for treating this orphan disease in children in this environment of rapidly changing medical practice.

This study is part of a Paediatric Investigational Plan (PIP; EMEA-000434-PIP01-08) agreed with the European Medicines Agency's Paediatric Committee (PDCO).

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PAH (WHO Group 1) with WHO class II or III symptoms in one of the following categories: Idiopathic, Heritable [familial], Secondary to connective tissue disease (e.g., limited scleroderma, diffuse scleroderma, mixed connective tissue disease (CTD), systemic lupus erythematosus, or overlap syndrome), or Persistent PAH despite surgical repair (at least 6 months prior to the screening visit) of atrial septal defects, ventricular septal defects, atrio-ventricular septal defects, and persistent patent ductus.
* Have met the following hemodynamic criteria for subjects with right heart catheterization (RHC) when performed as part of the diagnosis or routine care: mean pulmonary arterial pressure (mPAP) of >/=25 mmHg, pulmonary vascular resistance (PVR) of >/=240 dyne sec/cm5, left ventricular end diastolic pressure (LEVDP) or pulmonary capillary wedge pressure (PCWP) of ≤15 mmHg.
* be treatment naïve, have discontinued treatment with another ERA (e.g., bosentan) at least 1 month previously because of elevated liver function tests (LFTs), or have been on a stable dose of drug therapy for PAH (e.g., sildenafil or prostacyclin) for at least one month prior to the Screening Visit.
* Subjects who discontinued ERA treatment due to elevated LFTs, must have LFTs of <3 x Upper Limit of Normal (ULN).
* A female is eligible to participate in this study, as assessed by the investigator, if she is of: a. non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or, b. Child-bearing potential - has a negative pregnancy test and is not lactating at the Screening and Baseline/Randomisation Visits and, if sexually active, agrees to use 2 reliable methods of contraception from the Screening Visit until study completion and for at least 30 days following the last dose of study drug.
* Subject or subject's legal guardian is able and willing to give written informed consent. As part of the consent, female subjects of childbearing potential will be informed of the risk of teratogenicity and will need to be counselled in a developmentally appropriate manner on the importance of pregnancy prevention; and male subjects will need to be informed of potential risk of testicular tubular atrophy and aspermia.

Exclusion Criteria:

* currently taking an ERA.
* currently taking cyclosporine A.
* body weight is less than 20 Kg.
* have not tolerated PAH therapy due to adverse effects which may be related to their mechanism of action (e.g., prostanoids, ERA, PDE-5 inhibitors) with the exception of liver abnormalities for those subjects who were receiving another ERA.
* pregnant or breastfeeding.
* diagnosis of active hepatitis (hepatitis B surface antigen and hepatitis C antibody), or clinically significant hepatic enzyme elevation (i.e., ALT, AST or AP >3xULN) at Screening.
* severe renal impairment (creatinine clearance <30 mL/min) at Screening.
* clinically significant fluid retention in the opinion of the investigator.
* clinically significant anaemia in the opinion of the investigator.
* a known hypersensitivity to the study drug, the metabolites, or formulation excipients.
* have participated in another trial or have taken another investigational product during the previous 30 days.
* alcohol abuse, illicit drug use within 1 year.
* any concurrent condition or concurrent use of medication that would affect subject safety in the opinion of the investigator.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2013-11-12 (Actual); Study Completion 2013-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (4):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, New York, New York
- Argentina (3):
  - GSK Investigational Site, Guymallen, Mendoza Province
  - GSK Investigational Site, Ciudad de Buenos Aires
  - GSK Investigational Site, Córdoba
- France (3):
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Toulouse
- Germany (3):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Budapest, Hungary
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, San Donato Milanese (MI), Lombardy
- Japan (3):
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Russia (3):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
- GSK Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Ivy D, Beghetti M, Juaneda-Simian E, Miller D, Lukas MA, Ioannou C, Okour M, Narita J, Berger RMF. A Randomized Study of Safety and Efficacy of Two Doses of Ambrisentan to Treat Pulmonary Arterial Hypertension in Pediatric Patients Aged 8 Years up to 18 Years. J Pediatr X. 2020 Sep 22;5:100055. doi: 10.1016/j.ympdx.2020.100055. eCollection 2020 Spring. PMID 37332660
- [Derived] Okour M, Thapar MM, Farrell C, Lukas MA, Beghetti M, Beerahee M. Pediatric Population Pharmacokinetic Modeling and Exposure-Response Analysis of Ambrisentan in Pulmonary Arterial Hypertension and Comparison With Adult Data. J Clin Pharmacol. 2023 May;63(5):593-603. doi: 10.1002/jcph.2199. Epub 2023 Jan 29. PMID 36579617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the safety and efficacy of a high and low dose ambrisentan (adjusted as per participants body weight) administered orally in participants aged 8 to 18 years with pulmonary arterial hypertension (PAH).
Pre-assignment Details: A total of 41 participants were enrolled and randomized.
Groups:
- Low Dose Ambrisentan: Participants received ambrisentan low dose tablet either 2.5 milligram (mg) or 5 mg orally once daily for 24 weeks.
- High Dose Ambrisentan: Participants received ambrisentan high dose tablet either 5 mg, 7.5 mg or 10 mg orally once daily for 24 weeks.
Period: Overall Study
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Started | 21 | 20
Completed | 19 | 18
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Ambrisentan: Participants received ambrisentan low dose tablet either 2.5 mg or 5 mg orally once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.8 (2.70) | 12.3 (2.85) | 12.0 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 9 | 5 | 14
Race/Ethnicity, Customized [Number; unit: Count of participants]
  African American/African Heritage | 2 | 0 | 2
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - East Asian Heritage | 1 | 0 | 1
  Asian - Japanese Heritage | 5 | 0 | 5
  Asian - South East Asian Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 11 | 19 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Treatment-emergent Adverse Events (SAEs)
Description: AEs defined as any untoward medical occurrence in a patient or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAEs defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect, medical events that may not immediately life threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention as per medical or scientific judgement and events of drug-induced liver injury with hyperbilirubinaemia. Safety population comprised of all randomized participants who received at least 1 dose of study drug.
Time Frame: Up to 24 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Any AEs | 16 | 16
  Any SAEs | 6 | 2

2. Primary Outcome: Number of Participants With Post Baseline Potential Clinical Importance (PCI) Value for Clinical Chemistry Parameters: Alanine Amino Transferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT), Total Bilirubin and Creatinine
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: ALT, AST, GGT, total bilirubin and creatinine. PCI ranges were <3 times the upper limit of normal (ULN), <34.2 Micromoles per liter (UMOL/L) for total bilirubin and <176.8 (UMOL/L) for creatinine. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  ALT | 0 | 0
  AST | 0 | 0
  GGT | 0 | 0
  Total bilirubin | 1 | 0
  Creatinine | 0 | 0

3. Primary Outcome: Number of Participants With Post Baseline PCI Value for Hematology Parameter: Hemoglobin
Description: Blood samples were collected from participants for analysis of following hematology parameters: hemoglobin. PCI ranges were Males: 98 to180 grams per liter (G/L), Females: 91 to 161 (G/L) for hemoglobin. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Reference high range | 0 | 2
  Reference low range | 1 | 0

4. Primary Outcome: Number of Participants With Post Baseline PCI Value for Hematology Parameter: Hematocrit
Description: Blood samples were collected from participants for analysis of following hematology parameter: hematocrit. PCI ranges were males: <0.32 to >0.54, females: <0.29 to >0.506 proportion of red blood cells in blood for hematocrit. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Reference high range | 0 | 2
  Reference low range | 1 | 2

5. Primary Outcome: Number of Participants With Post Baseline PCI Value for Hematology Parameter: Platelet Count
Description: Blood samples were collected from participants for analysis of following hematology parameter: platelet count. PCI ranges were 100 to 400 for Giga cells per liter platelet count. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Reference high range | 0 | 0
  Reference low range | 0 | 1

6. Primary Outcome: Number of Participants With Abnormal Value for Physical Examination Parameter: Liver Size
Description: Physical examination included measurement of liver size. Any abnormal enlargement or reduction in the size of the liver is reported.
Time Frame: Week 12 and 24
Population: Safety population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Week 12, Abnormal: Improved, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Improved, n=20, 19 | 1 | 1
  Week 12, Abnormal: Worsened, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Worsened, n=20, 19 | 1 | 1
  Week 12, Abnormal: Unchanged, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Unchanged, n=20, 19 | 1 | 0
  Week 24, Abnormal: Improved, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Improved, n=19, 18 | 2 | 1
  Week 24, Abnormal: Worsened, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Worsened, n=19, 18 | 0 | 0
  Week 24, Abnormal: Unchanged, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Unchanged, n=19, 18 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Value for Physical Examination Parameter: Jugular Venous Pressure
Description: Physical examination of participants jugular venous pressure is measured.
Time Frame: Week 12 and 24
Population: Safety population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Week 12, Abnormal: Improved, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Improved, n=20, 19 | 0 | 1
  Week 12, Abnormal: Worsened, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Worsened, n=20, 19 | 0 | 1
  Week 12, Abnormal: Unchanged, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Unchanged, n=20, 19 | 0 | 3
  Week 24, Abnormal: Improved, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Improved, n=19, 18 | 0 | 1
  Week 24, Abnormal: Worsened, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Worsened, n=19, 18 | 1 | 0
  Week 24, Abnormal: Unchanged, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Unchanged, n=19, 18 | 0 | 4

8. Primary Outcome: Number of Participants With Abnormal Value for Physical Examination Parameter: Peripheral Edema
Description: Physical examination of paricipants peripheral edema is measured. Day 1 was considered as Baseline.
Time Frame: Week 12 and 24
Population: Safety population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Week 12, Abnormal: Improved, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Improved, n=20, 19 | 0 | 0
  Week 12, Abnormal: Worsened, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Worsened, n=20, 19 | 1 | 1
  Week 12, Abnormal: Unchanged, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Unchanged, n=20, 19 | 0 | 1
  Week 24, Abnormal: Improved, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Improved, n=19, 18 | 1 | 0
  Week 24, Abnormal: Worsened, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Worsened, n=19, 18 | 1 | 0
  Week 24, Abnormal: Unchanged, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Unchanged, n=19, 18 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal Value for Physical Examination Parameter: Ascites
Description: Physcial examination of paricipants ascites was measured. Day 1 was considered as Baseline.
Time Frame: Week 12 and 24
Population: Safety population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Week 12, Abnormal: Improved, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Improved, n=20, 19 | 0 | 0
  Week 12, Abnormal: Worsened, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Worsened, n=20, 19 | 0 | 0
  Week 12, Abnormal: Unchanged, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, Abnormal: Unchanged, n=20, 19 | 0 | 0
  Week 24, Abnormal: Improved, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Improved, n=19, 18 | 0 | 0
  Week 24, Abnormal: Worsened, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Worsened, n=19, 18 | 0 | 0
  Week 24, Abnormal: Unchanged, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, Abnormal: Unchanged, n=19, 18 | 0 | 0

10. Primary Outcome: Percentage of Physical Examination Parameter: Saturated Oxygen Level
Description: Physical examination of participants saturated oxygen level was measured. Day 1 was considered as Baseline.
Time Frame: Week 12 and 24
Population: Safety population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Percentage of oxygen saturation
  Week 12, n=20, 18: number analyzed (Participants) | 20 | 18
  Week 12, n=20, 18 | 96.9 (2.59) | 96.9 (6.93)
  Week 24, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, n=19, 18 | 97.3 (1.85) | 97.4 (1.92)

11. Primary Outcome: Number of Participants With Post Baseline PCI Value for Vital Signs Parameter: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. PCI ranges were <80 to >160 millimeters of mercury (mmHg) for SDP and <40 to >110 mmHg for DBP. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  SBP, Reference range high | 0 | 0
  SBP, Reference range low | 1 | 2
  DBP, Reference range high | 0 | 0
  DBP, Reference range low | 0 | 0

12. Primary Outcome: Number of Participants With Post Baseline PCI Value for Vital Signs Parameter: Heart Rate
Description: Heart rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. PCI ranges were <50 to >120 beats per minute (beats/min). Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Reference range high | 2 | 2
  Reference range low | 1 | 0

13. Primary Outcome: Number of Participants With Post Baseline PCI Value for Vital Signs Parameter: Weight
Description: Weight of the participants was measured. PCI ranges were <20 kilogram (kg) for weight. Only those parameters having any time post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to 24 Weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Participants
  Reference range high | 0 | 0
  Reference range low | 0 | 0

14. Primary Outcome: Change From Baseline of Pubertal Development: Men- Testicular Volume (TV) at Weeks 12 and 24
Description: Testicular volume was assessed by Prader's orchiodometer and the assessment was performed by a pediatric endocrinologist using the Tanner's criteria. Only those parameters having status - overall were presented. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 12 and 24
Population: Safety population. Only those male participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 9 | 5
Milliliter
  Week 12, Right TV, n=7, 4: number analyzed (Participants) | 7 | 4
  Week 12, Right TV, n=7, 4 | 0.4 (1.27) | 0.3 (0.50)
  Week 12, Left TV, n=8, 5: number analyzed (Participants) | 8 | 5
  Week 12, Left TV, n=8, 5 | 0.0 (0.53) | 0.2 (0.45)
  Week 24, Right TV, n=6, 4: number analyzed (Participants) | 6 | 4
  Week 24, Right TV, n=6, 4 | 0.5 (1.38) | 0.1 (0.25)
  Week 24, Left TV, n=7, 5: number analyzed (Participants) | 7 | 5
  Week 24, Left TV, n=7, 5 | 1.4 (2.76) | 0.5 (1.50)

15. Primary Outcome: Change From Baseline in Plasma Endocrine Parameter - Female : Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) at Weeks 12 and 24
Description: FSH and LH level of participants were measured. Only those parameters having status - overall were presented. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 12 and 24
Population: Safety population. Only those female participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per Liter
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 12 | 15
International unit per Liter
  Week 12, FSH, n=11, 13: number analyzed (Participants) | 11 | 13
  Week 12, FSH, n=11, 13 | 0.586 (1.412) | -0.023 (2.104)
  Week 24, FSH, n=10, 12: number analyzed (Participants) | 10 | 12
  Week 24, FSH, n=10, 12 | 0.010 (1.390) | 1.542 (2.518)
  Week 12, LH, n=11, 13: number analyzed (Participants) | 11 | 13
  Week 12, LH, n=11, 13 | 0.39 (3.117) | -0.28 (6.881)
  Week 24, LH, n=11, 13: number analyzed (Participants) | 11 | 13
  Week 24, LH, n=11, 13 | -0.56 (1.192) | 1.15 (6.806)

16. Primary Outcome: Change From Baseline in Plasma Endocrine Parameter - Female : Inhibin B at Weeks 12 and 24
Description: Inhibin B level of participants were measured. Only those parameters having status - overall were presented. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 12 and 24
Population: Safety population. Only those female participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 12 | 15
Nanogram per liter
  Week 12, Right TV, n=9, 7: number analyzed (Participants) | 9 | 7
  Week 12, Right TV, n=9, 7 | 4.9 (10.03) | 1.7 (33.70)
  Week 24, Left TV, n=9, 7: number analyzed (Participants) | 9 | 7
  Week 24, Left TV, n=9, 7 | -5.2 (36.44) | 16.0 (37.96)

17. Primary Outcome: Change From Baseline in Plasma Endocrine Parameter - Female : Sex Hormone Binding Globulin at Weeks 12 and 24
Description: Sex hormone binding globulin level of participants were measured. Only those parameters having status - overall were presented. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 12 and 24
Population: Safety population. Only those female participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 12 | 15
Milliliter
  Week 12, Right TV, n=10, 9: number analyzed (Participants) | 10 | 9
  Week 12, Right TV, n=10, 9 | 1.3 (9.55) | 7.4 (18.91)
  Week 24, Left TV, n=10, 8: number analyzed (Participants) | 10 | 8
  Week 24, Left TV, n=10, 8 | -9.2 (13.62) | 3.1 (14.21)

18. Secondary Outcome: Change From Baseline in the 6 Minutes Walking Distance (6MWD) Test
Description: Participant's 6MWD data has been presented into three categories as overall, with oxygen use and without oxygen use. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. NA indicates that standard deviation could not be calculated for single participant. Intent-to-Treat (ITT) population consist of all randomized participants who received at least one dose of study drug.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: Intent-to-treat population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Meters
  Week 4, Overall, n=21, 18: number analyzed (Participants) | 21 | 18
  Week 4, Overall, n=21, 18 | 33.10 (66.979) | 24.96 (71.254)
  Week 4, With oxygen use, n=2, 1: number analyzed (Participants) | 2 | 1
  Week 4, With oxygen use, n=2, 1 | -16.00 (11.314) | 85.20 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 4, Without oxygen use, n=19, 17: number analyzed (Participants) | 19 | 17
  Week 4, Without oxygen use, n=19, 17 | 38.27 (68.421) | 21.41 (71.793)
  Week 8, Overall, n=20, 18: number analyzed (Participants) | 20 | 18
  Week 8, Overall, n=20, 18 | 23.84 (65.154) | 37.70 (74.339)
  Week 8, With oxygen use, n=2, 1: number analyzed (Participants) | 2 | 1
  Week 8, With oxygen use, n=2, 1 | -16.00 (22.627) | 81.10 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 8, Without oxygen use, n=18, 17: number analyzed (Participants) | 18 | 17
  Week 8, Without oxygen use, n=18, 17 | 28.26 (67.133) | 35.15 (75.809)
  Week 12, Overall, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 12, Overall, n=19, 18 | 29.51 (79.657) | 40.29 (69.137)
  Week 12, With oxygen use, n=2, 1: number analyzed (Participants) | 2 | 1
  Week 12, With oxygen use, n=2, 1 | -1.00 (65.054) | 75.40 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 12, Without oxygen use, n=17, 17: number analyzed (Participants) | 17 | 17
  Week 12, Without oxygen use, n=17, 17 | 33.09 (82.121) | 38.22 (70.690)
  Week 16, Overall, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 16, Overall, n=19, 18 | 22.31 (88.832) | 36.43 (78.220)
  Week 16, With oxygen use, n=2, 1: number analyzed (Participants) | 2 | 1
  Week 16, With oxygen use, n=2, 1 | -21.00 (57.983) | 65.40 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 16, Without oxygen use, n=17, 17: number analyzed (Participants) | 17 | 17
  Week 16, Without oxygen use, n=17, 17 | 27.41 (91.681) | 34.73 (80.282)
  Week 20, Overall, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 20, Overall, n=19, 18 | 48.49 (90.645) | 31.19 (71.209)
  Week 20, With oxygen use, n=3, 1: number analyzed (Participants) | 3 | 1
  Week 20, With oxygen use, n=3, 1 | -0.33 (43.753) | 73.20 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 20, Without oxygen use, n=16, 17: number analyzed (Participants) | 16 | 17
  Week 20, Without oxygen use, n=16, 17 | 57.64 (95.070) | 28.72 (72.600)
  Week 24, Overall, n=18, 18: number analyzed (Participants) | 18 | 18
  Week 24, Overall, n=18, 18 | 55.14 (102.182) | 26.25 (62.011)
  Week 24, With oxygen use, n=3, 1: number analyzed (Participants) | 3 | 1
  Week 24, With oxygen use, n=3, 1 | 43.00 (53.395) | 65.90 (NA) — NA indicated that standard deviation could not be calculated for single participant.
  Week 24, Without oxygen use, n=15, 17: number analyzed (Participants) | 15 | 17
  Week 24, Without oxygen use, n=15, 17 | 57.57 (110.605) | 23.92 (63.100)

19. Secondary Outcome: Time to the First Clinical Worsening of Pulmonary Arterial Hypertension (PAH)
Description: Time to clinical worsening of PAH is defined as the time from randomization to the first occurrence of death or placed for lung transplant, hospitalization due to PAH deterioration, addition or increased dose of other targeted PAH therapeutic agents like prostanoids and PDE-5 inhibitors) and/or atrial septostomy, other PAH related deterioration identified by increase in WHO functional class, deterioration in exercise testing and clinical signs or symptoms of right sided heart failure.
Time Frame: Up to Week 24
Population: Intent-to-treat population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 3 | 3
Days | 77.3 (62.56) | 71.7 (29.26)

20. Secondary Outcome: Change From Baseline in Subject Global Assessment to Week 24 Using the SF-10 Health Survey for Children
Description: Short-form 10 (SF-10) Health Survey for Children is a 10-item parent-completed health assessment that measures physical and psychosocial functioning for children ages five and over. Each item has either 4, 5 or 6 response choices with associated point systems. Two summary scores were calculated: a Physical Summary Score (PHS) and a Psychosocial Summary Score (PSS) with a range of 5 to 30 points for each 5-item score. This aggregated point score was then standardized and transformed to a norm-based scoring metric in accordance with the developer's algorithms using associated mean and standard deviation derived from 2006 sample data. This generated the final standardized norm-based scores for PHS (range -10.90 to 57.21) and for PSS (range 8.81 to 62.28), respectively. A higher value on each summary score indicates better functioning. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Scores on a scale
  Physical health summary, n=16, 15: number analyzed (Participants) | 16 | 15
  Physical health summary, n=16, 15 | 0.194 (11.7733) | 2.811 (13.1172)
  Psychosocial summary, n=16, 15: number analyzed (Participants) | 16 | 15
  Psychosocial summary, n=16, 15 | 0.725 (8.6431) | 0.412 (10.1331)

21. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class to Week 24
Description: PAH was classified by WHO functional class (FC) at specific time points. There were four WHO FC grades based on severity of PAH symptoms (Class I=none, Class IV=most severe). Grades were then mapped to numeric scale, for which scores ranged from 1 to 4 (Class I=1 and Class IV=4). Score at Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: Intent-to-treat population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Scores on a scale
  Week 4, n=21, 19: number analyzed (Participants) | 21 | 19
  Week 4, n=21, 19 | -0.1 (0.36) | -0.1 (0.23)
  Week 8, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 8, n=20, 19 | -0.1 (0.45) | -0.1 (0.40)
  Week 12, n=20, 19: number analyzed (Participants) | 20 | 19
  Week 12, n=20, 19 | -0.1 (0.45) | 0.0 (0.58)
  Week 16, n=20, 18: number analyzed (Participants) | 20 | 18
  Week 16, n=20, 18 | -0.2 (0.49) | -0.2 (0.38)
  Week 20, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 20, n=19, 18 | -0.2 (0.50) | -0.2 (0.38)
  Week 24, n=19, 18: number analyzed (Participants) | 19 | 18
  Week 24, n=19, 18 | -0.3 (0.56) | -0.2 (0.43)

22. Secondary Outcome: Ratio to Baseline in Plasma N-terminal Pro-B Type Natriuretic Peptide (NT-Pro BNP) Concentration at Week 24
Description: NT-Pro BNP plasma concentrations were determined at specific time points. Geometric mean and SD logs has been presented. Day 1 was considered as Baseline. Ratio to Baseline is expressed as percentage change from Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline, Week 12 and 24
Population: Intent-to-treat population. Only those participants with available data at the specified time points were analyzed.
Measure: Geometric Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
Number analyzed (Participants) | 21 | 20
Percentage Change
  Week 12, n=19, 17: number analyzed (Participants) | 19 | 17
  Week 12, n=19, 17 | -15.93 (0.895) | -12.43 (0.862)
  Week 24, n=18, 17: number analyzed (Participants) | 18 | 17
  Week 24, n=18, 17 | -30.91 (0.851) | -28.25 (1.179)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non serious AEs were collected from the start of study treatment up to 24 weeks
Description: Safety Population was used. Safety Population comprised of all randomized participants who received at least one dose of a study drug
Arm/Group | Low Dose Ambrisentan | High Dose Ambrisentan
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/21 | 2/20
Other Adverse Events (participants affected / at risk) | 16/21 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Ambrisentan (N=21) | High Dose Ambrisentan (N=20)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Ambrisentan (N=21) | High Dose Ambrisentan (N=20)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT01332331/SAP_000.pdf
  • Study Protocol (2011-02-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT01332331/Prot_001.pdf